CLINICAL TRIAL: NCT03860584
Title: Alleviation Of Metabolic Endotoxemia In Adults With Metabolic Syndrome With Milk Fat Globule Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Professor and Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018H0564
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Syndrome; Metabolic Endotoxemia
Keywords: metabolic endotoxemia; milk fat globule membrane; gut health; endotoxin; inflammation; obesity
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Obesity

STUDY DESIGN:
Intervention Model Description: 2-arm, double-blind, randomized controlled, crossover trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and key research personnel will be blinded between MFGM-enriched full-fat dairy milk (treatment) and milk with soy phospholipid/lecithin (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFGM-enriched full-fat dairy milk (Experimental): Participants in this arm will receive MFGM-enriched full-fat dairy milk (3 servings/d) that contains MFGM at 10% phospholipid (relative to total lipid content) delivering MFGM at ~10-times that in full-fat dairy milk.
  Interventions: Dietary Supplement: MFGM-enriched full-fat dairy milk
- Soy phospholipid/lecithin milk (Placebo Comparator): Participants in this arm will receive a matched dairy milk that instead contains soy phospholipid/lecithin.
  Interventions: Dietary Supplement: Soy phospholipid/lecithin milk

INTERVENTIONS:
Dietary Supplement: MFGM-enriched full-fat dairy milk — MetS adults with metabolic endotoxemia will be enrolled to complete a 2-arm, double-blind, randomized controlled, crossover trial to test the independent benefits of MFGM. For each 2-wk arm, they will receive MFGM-enriched full-fat dairy milk (3 servings/d) or a matched dairy milk that instead contains soy phospholipid/lecithin (control). Milks have been formulated with soy lecithin or MFGM at 10% phospholipid (relative to total lipid content). This delivers MFGM at ~10-times that in full-fat dairy milk, which reflects that consumers obtain MFGM from dairy foods other than whole milk.
  Arms: MFGM-enriched full-fat dairy milk
Dietary Supplement: Soy phospholipid/lecithin milk — MetS adults with metabolic endotoxemia will be enrolled to complete a 2-arm, double-blind, randomized controlled, crossover trial to test the independent benefits of MFGM. For each 2-wk arm, they will receive MFGM-enriched full-fat dairy milk (3 servings/d) or a matched dairy milk that instead contains soy phospholipid/lecithin (control). Milks have been formulated with soy lecithin or MFGM at 10% phospholipid (relative to total lipid content).
  Arms: Soy phospholipid/lecithin milk

SUMMARY:
Metabolic syndrome (MetS) adults (n = 24; 18-65 y) will be enrolled to complete a 2-arm, double-blind, randomized controlled, crossover trial. They will be randomized in 4-unit blocks to receive, for 13 d, a controlled diet with dairy milk (3.5% fat; 3 servings/d) enriched with milk fat globule membrane (MFGM, MEB) or a matched dairy milk that instead contains soy lecithin/phospholipid (control, COMP). All foods during each study period will be provided to ensure weight maintenance and to increase homogeneity of gut and host responses. Anthropometrics and blood pressure will be assessed at days 0, 7, and 13. Prior to (day 0) and after each 2-wk arm (day 13), a fasting blood sample will be collected to assess serum endotoxin and metabolic chemistries (glucose, lipids, insulin), and Toll-like receptor 4 /nuclear factor kappaB (TLR4/NFκB)-dependent genes from whole blood. A breath sample will be collected to assess the correlation analysis of plasma metabolic biomarkers. After the 2-week intervention, from fecal samples collected on day 13, the investigators will assess microbiota composition and function, short chain fatty acids (SCFA), and intestinal inflammatory markers (calprotectin, myeloperoxidase). On d 13, participants in the fasted state will receive a high-fat/high-glucose meal challenge to induce gut-derived endotoxin translocation. At 30-minute intervals for 3-hour, the investigators will evaluate circulating endotoxin, glucose, and insulin; TLR4/NFκB-dependent genes will be assessed from whole blood at 0 hour and 3-hour. Gut permeability probes will be co-administered with the test meal challenge, and 24-hour urine will be collected to assess gut barrier integrity. Participants will then undergo a 2-week washout prior to receiving the alternative treatment and completing all procedures in an identical manner.

DETAILED DESCRIPTION:
Background and hypothesis:

Our preclinical evidence shows that phospholipid-rich milk fat globule membrane (MFGM) attenuates lipopolysaccharide-induced increases in gut permeability and pro-inflammatory cytokines. MFGM also attenuates inflammation in association with a prebiotic and/or antimicrobial activity that modulates microbiota composition. Our central hypothesis is that MFGM-enriched dairy milk compared with a matched milk beverage containing soy lecithin (control) decreases metabolic endotoxemia and improves glucose tolerance in metabolic syndrome (MetS) adults by increasing gut barrier integrity in association with alleviating gut dysbiosis and inflammation.

Study Design:

The investigators will enroll male and female MetS adults (n = 24; 18-65 y) to complete a 2-arm, double-blind, randomized controlled, crossover trial. They will be randomized in 4-unit blocks to receive, for 14 days, a controlled diet with dairy milk (3.5% fat; 3 servings/d) enriched with MFGM-derived phospholipid or a matched dairy milk that instead contains coconut and palm oil (control). The investigators will provide all foods during each study period to ensure weight maintenance and to increase homogeneity of gut and host responses.

Subjects:

Participants will be recruited from Columbus, Ohio area. Participants having no history of liver or cardiovascular disease or cancer will be enrolled. They will have ≥3 established criteria for MetS: i) glucose (100-126 mg/dL), ii) waist circumference (>89 or >102 cm for F/M), iii) HDL-C (<50 or <40 mg/dL in F/M), iv) triglyceride >150 mg/dL, and iv) blood pressure >130/85 mmHg. Major exclusion criteria include: unstable body mass (±2 kg over prior 3-mo) vegetarian; food allergies or lactose intolerance; user of dietary supplements or probiotics (within past 1-mo); pregnancy, lactation, changes in birth control (within 6-month); any gastrointestinal disorders; chronic diarrhea; smoker; excess alcohol (>2 drinks/day); excess aerobic exercise (>7 h/week); recent antibiotic or anti-inflammatory agent use; blood pressure >140/90 mmHg.

Dietary Control:

The intervention will be performed in the Human Nutrition Metabolic Kitchen under the auspice of a registered dietitian (PI Bruno). In each 2-wk intervention, participants' diet will be rigorously controlled. All foods will be prepared, packaged, and provided every 3-4 days to supply a weight maintenance (i.e. eucaloric) diet. To assess compliance, participants will return MFGM/coconut/palm oil milk bottles for counting and any uneaten food portions for weighed measurement. Milk beverages will also be formulated to contain para-aminobenzoic acid (PABA; 80 mg/milk serving). Spot urine samples will be collected 4 times during each study arm coinciding when participants pick up test foods. Urinary PABA will be measured by spectrophotometry. Separate from this, participants will also keep food logs to document any dietary deviation. Diets will be standardized at 50-60% of energy from carbohydrate with low fiber intakes (~15 g/day) similar to Americans' diets to prevent potential masking of the benefits of MFGM, 15-20% from protein, and 25-30% from fat. Importantly, other than test beverages provided as part of the eucaloric diet, diets will be otherwise devoid of significant amounts of dairy foods, fermented products, and probiotics to prevent confounding effects.

Measurements:

Anthropometrics and blood pressure will be assessed at days 0, 7, and 13. Prior to (day 0), at day 7 and after each 2-wk arm (day 13), a fasting blood sample will be collected to assess serum endotoxin and metabolic chemistries (glucose, insulin, lipids (triglyceride, total and HDL cholesterol), and TLR4/NFκB-dependent genes from whole blood. A breath sample will be collected to assess the correlation analysis of plasma metabolic biomarkers. After the 2-week intervention, from fecal samples collected on day 13, the investigators will assess microbiota composition and function, SCFAs, and intestinal inflammatory markers (calprotectin, myeloperoxidase). During this period, participants will also record daily stool characteristics using a 7-point Bristol Stool scale. On day 13, participants in the fasted state will receive a high-fat/high-glucose meal challenge to induce gut-derived endotoxin translocation. At 30-minute intervals for 3 hours, the investigators will evaluate circulating endotoxin, glucose, and insulin; TLR4/NFκB-dependent genes will be assessed from whole blood at 0 hour and 3-hour. Gut permeability probes will be co-administered with the test meal challenge, and 24-hour urine will be collected to assess gut barrier integrity. Participants will then undergo a 2-week washout prior to receiving the alternative treatment and completing all procedures in an identical manner.

ELIGIBILITY:
Inclusion Criteria:

* Serum Glucose 100-126 mg/dl
* Waist C >89/102 cm; F/M
* Serum HDL-C: <50/40 mg/dl; F/M
* Serum triglyceride: >150 mg/dl
* Blood Pressure >130/85 mmHg

Exclusion Criteria:

* Unstable body mass (±2 kg over prior 3-mo)
* Vegetarian
* Food allergies or lactose intolerance
* User of dietary supplements or probiotics (within past 1-mo)
* Pregnancy, lactation, changes in birth control (within 6-mo)
* Any gastrointestinal disorders
* Chronic diarrhea
* Smoker
* Excess alcohol (>2 drinks/d)
* Excess aerobic exercise (>5 h/wk)
* Recent antibiotic or anti-inflammatory agent use
* Blood Pressure >140/90 mmHg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pokala A, Kraft J, Taormina VM, Michalski MC, Vors C, Torres-Gonzalez M, Bruno RS. Whole milk dairy foods and cardiometabolic health: dairy fat and beyond. Nutr Res. 2024 Jun;126:99-122. doi: 10.1016/j.nutres.2024.03.010. Epub 2024 Mar 21. PMID 38669850
- [Background] Bruno RS, Pokala A, Torres-Gonzalez M, Blesso CN. Cardiometabolic health benefits of dairy-milk polar lipids. Nutr Rev. 2021 Dec 8;79(Suppl 2):16-35. doi: 10.1093/nutrit/nuab085. PMID 34879146
- [Background] Quarles WR, Pokala A, Shaw EL, Ortega-Anaya J, Hillmann L, Jimenez-Flores R, Bruno RS. Alleviation of Metabolic Endotoxemia by Milk Fat Globule Membrane: Rationale, Design, and Methods of a Double-Blind, Randomized, Controlled, Crossover Dietary Intervention in Adults with Metabolic Syndrome. Curr Dev Nutr. 2020 Jul 25;4(9):nzaa130. doi: 10.1093/cdn/nzaa130. eCollection 2020 Sep. PMID 32885133
- [Result] Pokala A, Quarles WR, Ortega-Anaya J, Jimenez-Flores R, Cao S, Zeng M, Hodges JK, Bruno RS. Milk-Fat-Globule-Membrane-Enriched Dairy Milk Compared with a Soy-Lecithin-Enriched Beverage Did Not Adversely Affect Endotoxemia or Biomarkers of Gut Barrier Function and Cardiometabolic Risk in Adults with Metabolic Syndrome: A Randomized Controlled Crossover Trial. Nutrients. 2023 Jul 23;15(14):3259. doi: 10.3390/nu15143259. PMID 37513677

RESULTS

PARTICIPANT FLOW:
Groups:
- MFGM Enriched Full-fat Dairy Milk Then Soy Phospholipid/Lecithin Milk: Participants in this sequence first received Milk fat globule membrane (MFGM) enriched full-fat dairy milk (3 servings/day for 2 weeks), followed by a 2-week washout, and then soy phospholipid/lecithin milk (3 servings/day for 2 weeks).
- Soy Phospholipid/Lecithin Milk Then MFGM-enriched Full-fat Dairy Milk: Participants in this sequence first received soy phospholipid/lecithin milk (3 servings/day for 2 weeks), followed by a 2-week washout, and then MFGM-enriched full-fat dairy milk (3 servings/day for 2 weeks).
Period: First Intervention (2 Weeks)
Arm/Group | MFGM Enriched Full-fat Dairy Milk Then Soy Phospholipid/Lecithin Milk | Soy Phospholipid/Lecithin Milk Then MFGM-enriched Full-fat Dairy Milk
Started | 17 | 13
Completed | 16 | 12
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | MFGM Enriched Full-fat Dairy Milk Then Soy Phospholipid/Lecithin Milk | Soy Phospholipid/Lecithin Milk Then MFGM-enriched Full-fat Dairy Milk
Started | 16 | 12
Completed | 16 | 12
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | MFGM Enriched Full-fat Dairy Milk Then Soy Phospholipid/Lecithin Milk | Soy Phospholipid/Lecithin Milk Then MFGM-enriched Full-fat Dairy Milk
Started | 16 | 12
Completed | 13 | 11
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Baseline characteristics of Metabolic Syndrome (MetS) participants at screening
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (5.5)
Waist circumference (cm) [Mean (Standard Deviation); unit: cm] | 102.1 (12.1)
Systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 121.0 (15.2)
Diastolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 81.5 (10.4)
Plasma Triglyceride (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 108.6 (95.6)
Plasma HDL-C (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 42.3 (13.7)
Plasma glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 99.7 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Serum Endotoxin
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: EU/ml
Groups:
- MFGM-enriched Full-fat Dairy Milk: Participants in this sequence first received MFGM-enriched full-fat dairy milk (3 servings/day for 2 weeks), followed by a 2-week washout, and then soy phospholipid/lecithin milk (3 servings/day for 2 weeks).
- Soy Phospholipid/Lecithin Milk: Participants in this sequence first received soy phospholipid/lecithin milk (3 servings/day for 2 weeks), followed by a 2-week washout, and then MFGM-enriched full-fat dairy milk (3 servings/day for 2 weeks).
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
EU/ml | 32.5 (2.3) | 30.6 (2.1)

2. Primary Outcome: Serum Endotoxin
Description: Data are biomarker area under the time-concentration curve (0-3 hours) on day 13
Time Frame: Day 13 (0, 30, 60, 90, 120, 150, 180 minutes post-meal challenge)
Measure: Mean (Standard Error); unit: EU/ml x min
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
EU/ml x min | 3855.4 (498.1) | 3972.6 (470.8)

3. Secondary Outcome: Plasma Glucose
Description: Data are biomarker area under the time-concentration curve (0-3 hours) on day 13
Time Frame: Day 13 (0, 30, 60, 90, 120, 150, 180 minutes post-meal challenge)
Measure: Mean (Standard Error); unit: mg/dL x min
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
mg/dL x min | 5453.6 (479.9) | 2124.1 (723.8)

4. Secondary Outcome: Plasma Glucose
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
mg/dL | 98.1 (1.6) | 99.6 (2.5)

5. Secondary Outcome: Plasma Insulin
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
uIU/mL | 15.1 (6.5) | 14.5 (6.0)

6. Secondary Outcome: Plasma Insulin
Description: Data are biomarker area under the time-concentration curve (0-3 hours) on day 13
Time Frame: day 13 (0, 30, 60, 90, 120, 150, 180 minutes post-meal challenge)
Measure: Mean (Standard Error); unit: uIU/mL x min
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
uIU/mL x min | 16253.2 (2017.0) | 13678.3 (1766.0)

7. Secondary Outcome: Plasma HDL-C
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
mg/dL | 32.3 (1.3) | 34.1 (1.4)

8. Secondary Outcome: Plasma Triglyceride
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
mg/dL | 101.7 (8.0) | 103.3 (9.9)

9. Secondary Outcome: Plasma Total Cholesterol
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
mg/dL | 187.0 (8.9) | 161.8 (8.3)

10. Secondary Outcome: Plasma Glucagon-like Peptide-1
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
pmol/L | 6.0 (1.6) | 6.7 (2.2)

11. Secondary Outcome: Urine Lactulose/Mannitol
Description: Data are the 24-hour urinary excretion ratio of lactulose relative to mannitol post-meal challenge on day 13
Time Frame: Day 13
Measure: Mean (Standard Error); unit: ratio
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
ratio | 0.0854 (0.0084) | 0.0777 (0.0069)

12. Secondary Outcome: Urine Sucralose/Erythritol
Description: Data are the 24-hour urinary excretion ratio of sucralose relative to erythritol post-meal challenge on day 13
Time Frame: 5-24 hours
Measure: Mean (Standard Error); unit: ratio
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
ratio | 0.0174 (0.0017) | 0.0172 (0.0014)

13. Secondary Outcome: Fecal Acetate
Description: Data are biomarker fecal concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
umol/g | 39.7 (3.5) | 42.1 (3.9)

14. Secondary Outcome: Fecal Butyrate
Description: Data are biomarker fecal concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
umol/g | 16.51 (1.81) | 19.96 (2.23)

15. Secondary Outcome: Fecal Propionate
Description: Data are biomarker fecal concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
umol/g | 21.38 (1.92) | 23.73 (2.71)

16. Secondary Outcome: Plasma Gastric Inhibitory Polypeptide
Description: Data are biomarker fasting concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
pg/mL | 67.0 (6.9) | 90.6 (13.2)

17. Secondary Outcome: Fecal Calprotectin
Description: Data are biomarker fecal concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: ug/g
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
ug/g | 47.8 (10.4) | 53.0 (13.3)

18. Secondary Outcome: Fecal Myeloperoxidase
Description: Data are biomarker fecal concentrations
Time Frame: Day 13
Measure: Mean (Standard Error); unit: ng/g
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
ng/g | 166.7 (18.4) | 163.6 (20.4)

19. Secondary Outcome: Whole-blood Messenger RNA Expression of Toll-like Receptor-4 at Fasting
Description: Data are expression levels of whole blood target gene normalized to housekeeping gene (β-actin) expression levels.
Time Frame: Day 13
Measure: Mean (Standard Error); unit: log2(fold change)
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
log2(fold change) | .087 (.06) | .91 (.07)

20. Secondary Outcome: Whole-blood Messenger RNA Expression of Interleukin-6 at Fasting
Description: Data are expression levels of whole blood target gene normalized to housekeeping gene (β-actin) expression levels.
Time Frame: Day 13
Measure: Mean (Standard Error); unit: log2(fold change)
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
log2(fold change) | 0.81 (0.11) | 0.71 (.15)

21. Secondary Outcome: Whole Blood Messenger RNA Expression of Tumor Necrosis Factor-alpha at Fasting
Description: Data are expression levels of whole blood target gene normalized to housekeeping gene (β-actin) expression levels.
Time Frame: Day 13
Measure: Mean (Standard Error); unit: log2(fold change)
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
log2(fold change) | 0.91 (0.10) | 0.83 (0.12)

22. Secondary Outcome: Whole Blood Messenger RNA Expression of Toll-like Receptor-4 at 3 h Post-meal Challenge
Description: Data are expression levels of whole blood target gene normalized to housekeeping gene (β-actin) expression levels measure at 3-hours post-meal challenge
Time Frame: Day 13, 3 h post-meal
Measure: Mean (Standard Error); unit: log2(fold change)
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
log2(fold change) | 0.89 (0.07) | 0.93 (0.07)

23. Secondary Outcome: Whole Blood Messenger RNA Expression of Interleukin-6 at 3 h Post-meal Challenge
Description: as for outcome 22
Time Frame: Day 13, 3 h post-meal
Measure: Mean (Standard Error); unit: log2(fold change)
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
log2(fold change) | 0.91 (0.12) | 0.85 (0.14)

24. Secondary Outcome: Whole Blood Messenger RNA Expression of Tumor Necrosis Factor-alpha at 3 h Post-meal Challenge
Description: as for outcome 22
Time Frame: Day 13, 3 h post-meal
Measure: Mean (Standard Error); unit: log2(fold change)
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
Number analyzed (Participants) | 24 | 24
log2(fold change) | 0.75 (0.07) | 0.97 (0.11)

ADVERSE EVENTS:
Time Frame: 3-months
Groups:
- MFGM-enriched Full-fat Dairy Milk: MetS adults with metabolic endotoxemia will be enrolled to complete a 2-arm, double-blind, randomized controlled, crossover trial to test the independent benefits of MFGM. For each 2-wk arm, they will receive either MFGM-enriched full-fat dairy milk (3 servings/d) or a matched dairy milk containing soy phospholipids/lecithin (control). Milks have been formulated with soy lecithin or MFGM at 10% phospholipid (relative to total lipid content).
- Soy Phospholipid/Lecithin Milk: MetS adults with metabolic endotoxemia will be enrolled to complete a 2-arm, double-blind, randomized controlled, crossover trial to test the independent benefits of MFGM. For each 2-wk arm, they will receive either MFGM-enriched full-fat dairy milk (3 servings/d) or a matched dairy milk containing soy phospholipids/lecithin (control).
Arm/Group | MFGM-enriched Full-fat Dairy Milk | Soy Phospholipid/Lecithin Milk
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03860584/Prot_SAP_000.pdf